CLINICAL TRIAL: NCT04750239
Title: Safety and Clinical Activity of Nivatrotamab, an Anti GD2×CD3 Bispecific Antibody, in Relapsed/Recurrent Metastatic Small-cell Lung Cancer An Open-label, Single-arm, Multicenter, Phase 1/2 Trial
Brief Title: Safety and Clinical Activity of Nivatrotamab in Relapsed/Recurrent Metastatic Small-cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to business priorities
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 402
Record Dates: First submitted 2021-02-06; First posted 2021-02-11 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-06

CONDITIONS: SCLC

STUDY DESIGN:
Intervention Model Description: open-label, single-arm, dose-escalation and expansion consisting of up to 13 cycles
Masking Description: open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivatrotamab (Experimental): Subcutaneous administration of nivatrotamab up to 13 cycles
  Interventions: Drug: Nivatrotamab

INTERVENTIONS:
Drug: Nivatrotamab — Anti GD2×CD3 monoclonal bi-specific antibody

SUMMARY:
Adult patients with small-cell lung cancer (SCLC) will be treated with nivatrotamab a monoclonal anti GD2×CD3 bispecific antibody to investigate the safety and tolerability of the drug.

DETAILED DESCRIPTION:
The study will include a phase 1 dose escalation part to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D). This will be conducted following a modified Bayesian Optimal Interval Design (mBOIN) design. For the purpose of dose escalation, dose-limiting toxicities (DLTs) will be collected and assessed for a period of 28 days (the DLT evaluation period).

A phase 2 dose expansion part will follow the phase 1 dose escalation. In phase 2, patients will be stratified according to whether they have platinum sensitive or platinum-resistant SCLC. Phase 2 will assess the long term safety and tolerability of nivatrotamab as well as the clinical activity of nivatrotamab when administered at the obtained MTD/RP2D in phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent has been provided prior to any trial-related procedures.
* Patient willing and able to comply with the trial protocol
* Age ≥18 years at the time of informed consent
* Histologically or cytologically proven SCLC. Radiographical relapse/progression after minimum 1 line of platinum-containing chemotherapy with partial response or complete response as the best response (only applicable for phase 2) and not more than 3 prior lines of therapy
* Measurable disease according to RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Expected survival >3 months
* Platelet counts ≥100,000 cells/mm3
* Hemoglobin ≥9 g/dL
* Absolute neutrophil count (ANC) ≥1000 cells/mm3
* Adequate liver function defined by aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≤3 × upper limit of normal (ULN), and serum bilirubin ≤1.5 × ULN with the following exceptions
* In patients with documented liver metastases, AST, ALT, and ALP ≤5 × ULN and serum bilirubin ≤1.5 × ULN
* Adequate renal function with serum creatinine ≤1.5 mg/dL or creatinine clearance ≥50 mL/min as calculated using the Cockcroft Gault equation
* Serum albumin >3.0 g/dL
* Women of child-bearing potential must agree to appropriate contraception during treatment and for a period of 30 days after the last dose of study drug.

Exclusion Criteria:

* Systemic chemotherapy, radiotherapy, immunotherapy, or major surgery administered within 3 weeks prior to the first planned dosing of the investigational Medicinal Product (IMP) per protocol
* Patients receiving any other investigational therapy for their cancer within 3 weeks prior to the first planned dosing of the IMP per protocol
* Patients who never received platinum-containing regimen for SCLC (defined as less than 2 cycles of platinum doublet)
* Persistent > grade 1 toxicity from previous treatment with checkpoint inhibitors
* Any immunosuppressive concomitant medication (i.e., salazopyrine, methotrexate, steroids etc.)
* Inability to wean off steroid, unless tapered to 0 mg/day minimum 10 days prior to the first treatment in case of prior use
* Any active, uncontrolled viral, fungal, or bacterial infection
* Any medical history within 3 months prior to enrolment with need for anticonvulsant therapy
* Patients with diagnosis of autoimmune diseases or immunodeficiencies or documented infection with human immunodeficiency virus (HIV) or hepatitis B or C virus (active)
* Previous autologous stem cell transplantation or solid organ transplantation
* Active heart disease including myocardial infarction within the last 6 months before first dose. This includes cardiac insufficiency with left ventricular ejection fraction (LVEF) <50%
* Active CNS metastases. Patients with treated central nervous system (CNS) metastases are eligible if they are clinically stable without any new neurological symptoms and if there is no radiological evidence of new or enlarging CNS metastases. CNS-directed treatment (surgery, radiation) must be completed 4 weeks prior to the first IMP administration.

Furthermore, patients are excluded if they have:

Leptomeningeal carcinomatosis Uncontrolled seizures. Patients with known seizure are eligible if they are stable and have been without seizure 4 weeks prior to the first IMP administration

* Patients who experienced severe or recurrent (>grade 2) immune mediated adverse events (AEs) or infusion related reactions (IRRs), including those that lead to permanent discontinuation while on treatment with immune oncology agents
* Prior treatment with anti-GD2 antibody or bispecific antibodies
* Patients with Limited Disease (LD), who are candidates for local or regional therapy.
* Impending need for palliative radiotherapy or surgery for pathological fractures and/or for medullary compression up to 3 weeks prior to the first planned dosing of the IMP per protocol (palliative radiation for other reasons within 2 weeks)
* History of other active malignancy within the past 3 years prior to the first planned dosing of the IMP per protocol (excluding non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, incidental prostate cancer (T1a, Gleason score ≤ 6, prostate specific antigen (PSA) less than 0.5 ng/ml)
* Patients with a significant intercurrent illness (any ongoing serious medical problem unrelated to cancer or its treatment) that is not covered by the detailed exclusion criteria and that is expected to interfere with the action of the trial IMP or significantly increase the severity of the toxicities experienced from trial treatment
* Patients who are pregnant or breastfeeding
* Patients with a body weight of < 45 kg
* Patients with prior orthostatic hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivatrotamab 50 mcg (Dose Level 1): Subcutaneous administration of nivatrotamab up to 13 cycles
  Nivatrotamab: Anti GD2×CD3 monoclonal bi-specific antibody
Period: Overall Study
Arm/Group | Nivatrotamab 50 mcg (Dose Level 1)
Started | 3
Completed | 0
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Trial terminated by sponsor | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Arm/Group | Nivatrotamab 50 mcg (Dose Level 1)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 66.0 [64 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLTs) Phase I
Description: Summary of DLTs in DLT evaluable subjects.
Time Frame: Days 1 through 28
Population: DLT Evaluable Analysis Set
Measure: Number; unit: participants
Arm/Group | Nivatrotamab 50 mcg (Dose Level 1)
Number analyzed (Participants) | 2
participants | 1

2. Primary Outcome: Number of Participants With Adverse Events (AEs) for Different Doses of Nivatrotamab in Phase I
Description: Number of participants with adverse events as a measure of safety and tolerability.
Time Frame: From first dose until 30 days after last IMP, up to 26 weeks. Actual duration for treated patients were from 21 to 58 days.
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Nivatrotamab 50 mcg (Dose Level 1): Nivatrotamab dose level 50 mcg
Arm/Group | Nivatrotamab 50 mcg (Dose Level 1)
Number analyzed (Participants) | 3
Participants
  Any Adverse Event | 3
  Any Serious Adverse Event | 3

ADVERSE EVENTS:
Time Frame: From first dose until 30 days after last IMP, up to 26 weeks. Actual duration for treated patients were from 21 to 58 days.
Description: Non-serious AEs were reported from the day of the first IMP administration until 30 days after the last IMP administration.
Arm/Group | Nivatrotamab 50 mcg (Dose Level 1)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivatrotamab 50 mcg (Dose Level 1) (N=3)
Cytokine release syndrome (Immune system disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivatrotamab 50 mcg (Dose Level 1) (N=3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Herpes simplex (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated after 3 subjects due to a business strategy decision. At this point the maximum tolerated dose was not established. Only 3 subjects at dose level 1 (nivatrotamab 50 mcg) were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT04750239/Prot_SAP_000.pdf